CLINICAL TRIAL: NCT01976858
Title: A Double-Blind, Multicenter, Randomized Study Evaluating the Safety, Tolerability and Pharmacokinetic/Pharmacodynamic Relationship in T2DMs Treated With 8 Weeks Injection of Polyethylene Glycol Loxenatide
Brief Title: A Phase I Study of 8-week Continuous Treatment With Polyethylene Glycol Loxenatide in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEX168-I-03
Record Dates: First submitted 2013-10-22; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: PEX168, diabetes, phase I
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — polyethylene glycol loxenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PEX168 50 microgram (Experimental): PEX168 50 microgram qw sc. and the medication continued for 8 weeks
  Interventions: Drug: PEX168
- PEX168 100 microgram (Experimental): PEX168 100 microgram qw sc. and the medication continued for 8 weeks
  Interventions: Drug: PEX168
- PEX168 200 microgram (Experimental): PEX168 200 microgram qw sc. and the medication continued for 8 weeks
  Interventions: Drug: PEX168
- PEX168 300 microgram (Experimental): PEX168 300 microgram qw sc. and the medication continued for 8 weeks
  Interventions: Drug: PEX168
- Placebo (Placebo Comparator): Placebo qw sc. and the medication continued for 12 weeks
  Interventions: Drug: PEX168

INTERVENTIONS:
Drug: PEX168 — A injection administered subcutaneously
  Other Names: Polyethylene Glycol Loxenatide

SUMMARY:
Polyethylene Glycol Loxenatide (PEX168) is a new human glucagon-like peptide 1 (GLP-1) analogue that created on the basis of the Exenatide and modified by polyethylene glycol (PEG).

This study aims to evaluate the PK, PD and safety by 8-week continuous treatment of PEX168.

ELIGIBILITY:
Inclusion Criteria:

1. aged 20-65 years old, male or female, diagnosis of type 2 diabetes according to the 1999 WHO criteria more than 3 months.
2. HbA1C 7.0-10.0% and fasting plasma glucose 7.0-10.0 mmol/L after treatment of diet, exercise or a single oral hypoglycemic agents (metformin , glimepiride or pioglitazone).
3. unused insulin within 3 months prior to the enrollment.
4. Body mass index within the range from 19 to 35, and body weight does not changes exceeding 10% in the past 3 months.
5. Normol liver, kidney, heart function.
6. Willing to use physical means of contraception during the trial stage.
7. voluntarily to participate in the study.

Exclusion Criteria:

1. 1 diabetes.
2. used GLP-1, GLP-1 analogs or DPP-4 inhibitors in the past 3 months.
3. have diabetic ketoacidosis , diabetic hyperosmolar nonketotic coma patients with a history
4. There is a history of severe hypoglycemia : such as low blood sugar cause drowsiness , unconsciousness , nonsense , and even coma.
5. with severe diabetes complications ( renal , retinal , nerve , vascular disease).
6. has acute and chronic pancreatitis history ;
7. heart failure , unstable angina , severe arrhythmia, patients with a history of myocardial infarction ;
8. There is a history of hypertension and blood pressure is not well controlled : SBP> 160mmHg and / or DBP> 95mmHg persons ;
9. severe chronic gastrointestinal disease ( active ulcer nearly six months ) or have been affecting drug absorption in patients treated ;
10. There are obvious blood system diseases ;
11. There are other endocrine system diseases , such as hyperthyroidism , etc. ;
12. with severe trauma or surgery , severe infection ;
13. have mental illness , drug or other substance abuse or alcoholism ( drinking at least 2 times per week , more than 100g each drink ) ;
14. used any drugs that may affect the study , within 3 months before treatment as the subjects participated in any clinical trials ;
15. within the past six months more than 400ml of blood loss (including blood , trauma or other reasons ) ;
16. were receiving steroids or are receiving cancer treatment ;
17. has been prepared during pregnancy or pregnancy test in female patients ;
18. hepatitis B HBeAg , hepatitis C antibody positive , HIV antibody positive , syphilis antibody positive .
19. skin test positive of PEX168;
20. The researchers considered any factors that the subject should not participate in this trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine serum concentrations of PEX168 | 8 weeks

SECONDARY OUTCOMES:
To determin HbA1c levels of PEX168 | 8 weeks

OTHER OUTCOMES:
To assess number of participants with Adverse Events as a Measure of Safety and To assess number of participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jinkui Yang, Ph.D, M.D, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing tongren hospital, Beijing, Beijing Municipality, China